CLINICAL TRIAL: NCT07400068
Title: Effect of Adjunct Transforaminal Anterior Epidural Steroid Injection Following Percutaneous Laser Disc Decompression in Patients With Single-Level Lumbar Disc Herniation: A Prospective Observational Study
Brief Title: PLDD With or Without Transforaminal Epidural Steroid Injection in Lumbar Disc Herniation
Acronym: PLDD-TFESI
Status: Not yet recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mesut Bakır, Associate Professor of Anesthesiology and Algology, Mersin University
Other Study IDs: MU-PLDD-TFESI-2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Disc Herniation; Lumbar Radiculopathy
Keywords: Percutaneous Laser Disc Decompression; Transforaminal Epidural Steroid Injection; Minimally Invasive Spine Treatment; Radicular Pain; PLDD
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLDD Alone: Patients with single-level lumbar disc herniation who undergo routine percutaneous laser disc decompression (PLDD) as part of standard clinical care without adjunct epidural steroid injection.
  Interventions: Procedure: Percutaneous Laser Disc Decompression (PLDD)
- PLDD Plus Transforaminal Epidural Steroid Injection: Patients with single-level lumbar disc herniation who undergo routine percutaneous laser disc decompression (PLDD) followed by adjunct transforaminal anterior epidural steroid injection with dexamethasone during the same session as part of standard clinical care.
  Interventions: Procedure: Transforaminal Anterior Epidural Steroid Injection

INTERVENTIONS:
Procedure: Percutaneous Laser Disc Decompression (PLDD) — Routine minimally invasive laser-based disc decompression performed under fluoroscopic guidance to reduce intradiscal pressure in patients with lumbar disc herniation.
  Groups: PLDD Alone
Procedure: Transforaminal Anterior Epidural Steroid Injection — Routine transforaminal anterior epidural injection of dexamethasone performed under fluoroscopic guidance following PLDD during the same session without additional puncture.
  Groups: PLDD Plus Transforaminal Epidural Steroid Injection

SUMMARY:
This prospective observational study aims to evaluate the clinical outcomes of patients with single-level lumbar disc herniation who undergo routine percutaneous laser disc decompression (PLDD).

In routine clinical practice, some patients receive an additional transforaminal anterior epidural steroid injection during the same session without an extra puncture. This study will prospectively follow patients who receive PLDD alone and those who receive PLDD combined with epidural steroid injection.

Pain intensity, functional status, analgesic use, need for additional interventions, and complications will be assessed over time. The results may help to clarify whether adding epidural steroid injection to PLDD improves clinical outcomes in patients with lumbar disc herniation.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study conducted at the Algology Clinic of Mersin University Faculty of Medicine. The study will include adult patients with single-level lumbar disc herniation confirmed by magnetic resonance imaging who undergo routine percutaneous laser disc decompression (PLDD) as part of standard clinical care.

According to routine clinical practice and physician decision, some patients receive adjunct transforaminal anterior epidural steroid injection with dexamethasone in the same session following PLDD using the same cannula after withdrawal from the disc space and confirmation of epidural position with contrast under fluoroscopy. This combined approach does not require an additional puncture and is part of standard clinical treatment.

Patients will be prospectively followed and divided into two groups based on routine clinical management: those undergoing PLDD alone and those undergoing PLDD with adjunct transforaminal epidural steroid injection.

Baseline demographic data including age and sex, clinical characteristics such as symptom duration and affected disc level, and comorbidities will be recorded using standardized data collection forms.

The primary outcome measure will be change in leg pain intensity assessed by the Numeric Rating Scale (NRS). Secondary outcome measures will include back pain NRS, functional status evaluated using the Oswestry Disability Index (ODI), analgesic consumption, need for additional interventions, and complication rates.

Follow-up assessments will be conducted at baseline, 2 weeks, 6 weeks, 3 months, and 6 months after the procedure through outpatient visits or telephone interviews.

All procedures included in this study are part of routine clinical practice, and no experimental interventions will be performed. Data will be collected and analyzed in accordance with ethical standards and patient confidentiality.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years and older

Diagnosis of single-level lumbar disc herniation confirmed by magnetic resonance imaging (MRI)

Presence of radicular leg pain refractory to conservative treatment

Undergoing routine percutaneous laser disc decompression (PLDD) as part of standard clinical care

Ability to provide informed consent

Exclusion Criteria:

Multilevel lumbar disc herniation

Extruded or sequestered disc herniation

Severe spinal canal stenosis or spinal instability

Previous lumbar spine surgery at the affected level

Active infection or systemic inflammatory disease

Coagulopathy or use of anticoagulant therapy contraindicating intervention

Pregnancy

Inability to complete follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older with single-level lumbar disc herniation confirmed by magnetic resonance imaging who undergo routine percutaneous laser disc decompression at a tertiary university algology clinic will be included. Patients may receive PLDD alone or PLDD combined with adjunct transforaminal anterior epidural steroid injection according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Leg Pain Intensity (NRS) | Baseline to 1 month after procedure
  Change in leg pain intensity assessed using the Numeric Rating Scale (NRS, 0-10), where 0 indicates no pain and 10 indicates worst possible pain.

SECONDARY OUTCOMES:
Change in Back Pain Intensity (NRS) | Baseline to 1 month after procedure
  Change in low back pain intensity assessed using the Numeric Rating Scale (NRS, 0-10).
Functional Disability (Oswestry Disability Index) | Baseline to 1 month after procedure
  Functional status assessed using the Oswestry Disability Index (ODI), a validated questionnaire measuring disability related to low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Bakır, Principal Investigator — Mersin University Faculty of Medicine, Pain Clinic
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality considerations and institutional data protection policies. The collected data will be used solely for the purposes of this study and related scientific publications.

REFERENCES:
- [Background] Foresti ML, Ferreira ML. Lipase-catalyzed acidolysis of tripalmitin with capric acid in organic solvent medium: Analysis of the effect of experimental conditions through factorial design and analysis of multiple responses. Enzyme Microb Technol. 2010 May 5;46(6):419-29. doi: 10.1016/j.enzmictec.2010.01.002. Epub 2010 Jan 21. PMID 25919616
- [Background] Benyamin RM, Manchikanti L, Parr AT, Diwan S, Singh V, Falco FJ, Datta S, Abdi S, Hirsch JA. The effectiveness of lumbar interlaminar epidural injections in managing chronic low back and lower extremity pain. Pain Physician. 2012 Jul-Aug;15(4):E363-404. PMID 22828691
- [Background] Giger JM, Haddad F, Qin AX, Zeng M, Baldwin KM. Effect of unloading on type I myosin heavy chain gene regulation in rat soleus muscle. J Appl Physiol (1985). 2005 Apr;98(4):1185-94. doi: 10.1152/japplphysiol.01099.2004. Epub 2004 Dec 10. PMID 15591287